CLINICAL TRIAL: NCT04473430
Title: Study to Determine the Efficacy of Real-time CGM in Preventing Hypoglycemia Among Insulin-treated Patients With DM2 on Hemodialysis, Compared to Standard of Care (POC BG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rodolfo Galindo, Principal Investigator, Emory University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00114840; MH121653 (Other: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)); 1K23DK123384-01 (NIH)
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: End-Stage Renal Disease; Type 2 Diabetes
Keywords: ESRD; Continuous Glucose Monitoring; Diabetes
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Patients with type 2 DM treated with insulin and receiving hemodialysis will use a real-time/personal CGM for 4 weeks (Intervention-Control Group), then 2 weeks of wash-out period, and cross over to use POC BG for 4 weeks; and vice versa (Control-Intervention Group).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Real-time Dexcom CGM during CGM Intervention (Experimental): Patients with type 2 DM treated with insulin and receiving hemodialysis will use a real-time/personal CGM for 4 weeks (Intervention-Control Group), then 2 weeks of wash-out period, and cross over to use POC BG for 4 weeks, for insulin adjustments.
  Interventions: Device: Dexcom Real-time G6 Continuous Glucose Monitoring System (CGM)
- Professional Dexcom CGM During Point-Of-Care Blood Glucose Intervention (Experimental): Patients with type 2 DM treated with insulin and receiving hemodialysis will use POC BG for 4 weeks, then 2 weeks of wash-out period, and cross over to use a real-time/personal CGM for 4 weeks, for insulin adjustments (Control-Intervention Group).
  Interventions: Device: POC Glucose Testing

INTERVENTIONS:
Device: Dexcom Real-time G6 Continuous Glucose Monitoring System (CGM) — Dexcom G6, a factory-calibrated CGM system, is innovative in many aspects: 1) it does not require finger stick POC BG for calibration, 2) the sensor is small, compact, light-weight, 3) has no interference with several substance and drugs, and 4) protective "urgent low soon" alarm, with proven prediction of hypoglycemia within 20 minutes in advance.
  Dexcom G6 monitors glucose continuously (24 hrs) and displays real-time glucose values, glucose trends/arrows and alarms, including the "urgent low soon" alarm (predictive of hypoglycemia < 55 mg/dL within the preceding 20 minutes).
  Diagnostic Test: Real-time CGM will be used to collect outcomes variables
  Arms: Real-time Dexcom CGM during CGM Intervention
Device: POC Glucose Testing — POC BG (standard of care) uses commercially-available glucose meters for blood glucose monitoring. It is approved to be used in dialysis populations.
  Diagnostic Test: Professional CGM will be used to collect outcomes variables (including during the POC BG testing).
  Arms: Professional Dexcom CGM During Point-Of-Care Blood Glucose Intervention

SUMMARY:
The study is conducted to assess the efficacy of real-time CGM data in preventing hypoglycemia in patients with type 2 diabetes and end-stage kidney disease (ESKD), treated with insulin therapy and receiving hemodialysis.

DETAILED DESCRIPTION:
The study is conducted to assess the efficacy of real-time CGM data in preventing hypoglycemia among patients with type 2 diabetes (DM2), treated with insulin and receiving hemodialysis. The study will provide novel insights into the glycemic exposure patterns among dialysis patients and will provide preliminary data for future outcomes-based studies determining the best glycemic targets for this group.

ELIGIBILITY:
Inclusion Criteria:

* adult subjects with type 2 diabetes
* receiving hemodialysis (for at least 90 days)
* treated with insulin therapy [basal insulin alone (glargine U100, glargine U300, detemir, degludec, NPH)], or in combination with bolus insulin (at least one or more injections of aspart, lispro, glulisine, regular insulin) or in combination with incretin therapy (DPPIV or GLP1)
* willingness to wear the CGM
* currently performing self-monitored blood glucose (at least 2 times daily).

Exclusion Criteria:

* use of sulfonylureas or thiazolidinediones alone or in combination with insulin
* use of personal/real-time CGM 3 months prior to study entry (blinded CGM is allowed)
* prior use of insulin pumps or hybrid close loop systems (for at least the prior 28 days)
* current or anticipated use of stress steroids doses (prednisone ≤5mg or its equivalent is allowed)
* subjects who are sensitive or allergic to adhesive
* extensive skin changes/diseases that preclude wearing the required number of devices on normal skin (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites
* any condition that, in the opinion of the Investigator, would interfere with their participation in the trial (e.g., marked visual or hearing impairment, active alcohol or drug abuse, mental illness) or pose excessive risk to study staff handling venous blood samples
* situations that will limit the subject's ability to comply with the protocol (per investigator discretion)
* active malignancy
* unable to give informed consent
* at least 10% of time spent in clinical relevant hypoglycemia (<54 mg/dl) during blinded CGM period
* significant hypoglycemia (< 40 mg/dL)
* severe hyperglycemia (BG> 400 mg/dL)
* extensive skin abnormalities at insertion sites
* pregnancy or breastfeeding
* severe anemia (Hemoglobin < 5 mg/dl)
* polycythemia (Hemoglobin >17 mg/dl)
* subjects taking acetaminophen (more than 1 gr every six hours)
* hydroxyurea (may cause interference with the sensor membrane).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Clinic, Atlanta, Georgia
  - Grady Health System (non-CRN), Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared
Supporting Information: Study Protocol
Time Frame: Start 6 months after publication End 12 months after publication
Access Criteria: Researchers who provide a methodologically sound proposal to achieve the aims in the approved proposal will get access. Proposals should be directed to rodolfo.galindo@emory.edu.
  To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 66 individuals who signed the informed consent form (ICF), 53 took part in the study. The remaining 13 individuals did not proceed to the study due to screening failure. Therefore, the following tables include data only from the 53 participants who began the study.
Groups:
- Real-time Dexcom CGM During CGM Intervention, Then Professional Dexcom CGM During POC Intervention: Patients with type 2 DM treated with insulin and receiving hemodialysis will use a real-time/personal CGM for 4 weeks (Intervention-Control Group), then 2 weeks of wash-out period, and cross over to use POC BG for 4 weeks.
  Dexcom real-time G6 CGM System: Dexcom G6, a factory-calibrated CGM system, is innovative in many aspects: 1) it does not require finger stick POC BG for calibration, 2) the sensor is small, compact, light-weight, 3) has no interference with several substance and drugs, and 4) protective "urgent low soon" alarm, with proven prediction of hypoglycemia within 20 minutes in advance. It uses a novel semi-permeable membrane that blocks interference with most clinically relevant substances, including high levels of urea and creatinine, and commonly used medications. Dexcom G6 CGM is a commercially-available, minimally invasive sensor, with a flexible and thin wire that is inserted into the abdominal subcutaneous tissue. It monitors glucose continuously (24 hrs) and displays real-time glucose values, glucose trends/arrows and alarms, including the "urgent low soon" alarm (predictive of hypoglycemia < 55 mg/dL within the preceding 20 minutes).
  Diagnostic Test: Real-time CGM will be used to collect outcomes variables
- Professional Dexcom CGM During POC Intervention, Then Real-time Dexcom CGM During CGM Intervention: Patients with type 2 DM treated with insulin and receiving hemodialysis will use POC BG for 4 weeks, then 2 weeks of wash-out period, and cross over to use a real-time/personal CGM for 4 weeks (Control-Intervention Group).
  Intervention: POC BG (standard of care) uses commercially-available glucose meters for blood glucose monitoring. It is approved to be used in dialysis populations.
  Diagnostic Test: CGM will be used to collect outcomes variables during each phase (including during the POC BG testing).
Period: Phase I (First Intervention - 4 Weeks)
Arm/Group | Real-time Dexcom CGM During CGM Intervention, Then Professional Dexcom CGM During POC Intervention | Professional Dexcom CGM During POC Intervention, Then Real-time Dexcom CGM During CGM Intervention
Started | 25 | 28
Completed | 21 | 27
Not Completed | 4 | 1
Period: Phase II (Second Intervention - 4 Weeks)
Arm/Group | Real-time Dexcom CGM During CGM Intervention, Then Professional Dexcom CGM During POC Intervention | Professional Dexcom CGM During POC Intervention, Then Real-time Dexcom CGM During CGM Intervention
Started | 21 | 27
Excluded From Analysis ((Missing CGM data)) | 1 | 0
Completed | 17 | 23
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants received either Real-time Dexcom CGM Intervention or POC-BG Intervention first, and then switch to the remaining intervention after a 2 week wash out period.
  Participants will use either CGM or POC BG testing (during each assignment phase) for insulin adjustment. CGM will be used to collect outcomes variables during each phase (including during the POC BG testing).
Arm/Group | All Participants
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.36 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Differences in Mean Percentage Time-in-hypoglycemia (< 70 mg/dL)
Description: Differences in mean percentage time-in-hypoglycemia (< 70 mg/dL) during the intervention phase in both groups (i.e. Real-time Dexcom CGM During CGM Intervention vs. Professional Dexcom CGM During Point-of-Care Glucose Intervention), as measured by CGM.
  Participants will use either CGM or POC BG testing (during each assignment phase) for insulin adjustment. CGM will be used to collect outcomes variables during each phase (including during the POC BG testing).
Time Frame: 8 weeks (after completion of both phases)
Population: Population analyzed per group included patients with usable data.
Measure: Mean (Standard Deviation); unit: percentage of time in hypoglycemia
Groups:
- Real-time Dexcom CGM: Patients with type 2 DM treated with insulin and receiving hemodialysis will use a real-time/personal CGM for 4 weeks (Intervention-Control Group), then 2 weeks of wash-out period, and cross over to use POC BG for 4 weeks.
  Intervention: Dexcom real-time G6 Continuous Glucose Monitoring System (CGM): Dexcom G6, a factorycalibrated CGM system, is innovative in many aspects: 1) it does not require finger stick POC BG for calibration, 2) the sensor is small, compact, light-weight, 3) has no interference with several substance and drugs, and 4) protective "urgent low soon" alarm, with proven prediction of hypoglycemia within 20 minutes in advance. The sensor uses a novel semi-permeable membrane that blocks interference with most clinically relevant substances, including high levels of urea and creatinine, and commonly used medications. Dexcom G6 CGM is a commercially-available, minimally invasive sensor, with a flexible and thin wire that is inserted into the abdominal subcutaneous tissue. Dexcom G6 monitors glucose continuously (24 hrs) and displays realtime glucose values, glucose trends/arrows and alarms, including the "urgent low soon" alarm (predictive of hypoglycemia < 55 mg/dL within the preceding 20 minutes).
  Diagnostic Test: Real-time CGM will be used to collect outcomes variables
- Professional Dexcom CGM (Blinded): Patients with type 2 DM treated with insulin and receiving hemodialysis will use POC BG for 4 weeks, then 2 weeks of wash-out period, and cross over to use a real-time/personal CGM for 4 weeks.
  Intervention: POC BG (standard of care) uses commercially-available glucose meters for blood glucose monitoring. It is approved to be used in dialysis populations.
  Diagnostic Test: CGM will be used to collect outcomes variables during each phase (including during the POC BG testing).
Arm/Group | Real-time Dexcom CGM | Professional Dexcom CGM (Blinded)
Number analyzed (Participants) | 39 | 39
percentage of time in hypoglycemia | 1.24 (1.82) | 1.19 (2.79)

2. Secondary Outcome: % Time in Target Range (70-180 mg/dl)
Description: % time in target range (70-180 mg/dl) during the intervention phase in both groups (i.e. Real-time Dexcom CGM During CGM Intervention vs. Professional Dexcom CGM During Point-of-Care Glucose Intervention), as measured by CGM.
  Participants will use either CGM or POC BG testing (during each assignment phase) for insulin adjustment. CGM will be used to collect outcomes variables during each phase (including during the POC BG testing).
Time Frame: 8 weeks (after completion of both phases)
Population: Population analyzed per group included patients with usable data.
Measure: Mean (Standard Deviation); unit: percentage of time in target range
Groups:
- Real-time Dexcom CGM: Patients with type 2 DM treated with insulin and receiving hemodialysis will use a real-time/personal CGM for 4 weeks (Intervention-Control Group), then 2 weeks of wash-out period, and cross over to use POC BG for 4 weeks.
  Intervention: Dexcom real-time G6 Continuous Glucose Monitoring System (CGM): Dexcom G6, a factorycalibrated CGM system, is innovative in many aspects: 1) it does not require finger stick POC BG for calibration, 2) the sensor is small, compact, light-weight, 3) has no interference with several substance and drugs, and 4) protective "urgent low soon" alarm, with proven prediction of hypoglycemia within 20 minutes in advance. The sensor uses a novel semi-permeable membrane that blocks interference with most clinically relevant substances, including high levels of urea and creatinine, and commonly used medications. Dexcom G6 CGM is a commercially-available, minimally invasive sensor, with a flexible and thin wire that is inserted into the abdominal subcutaneous tissue. Dexcom G6 monitors glucose continuously (24 hrs) and displays realtime glucose values, glucose trends/arrows and alarms, including the "urgent low soon" alarm (predictive of hypoglycemia < 55 mg/dL within the preceding 20 minutes). POC BG: Real-time CGM will be used to collect outcomes variables
- Professional Dexcom CGM (Blinded): Patients with type 2 DM treated with insulin and receiving hemodialysis will use POC BG for 4 weeks, then 2 weeks of wash-out period, and cross over to use a real-time/personal CGM for 4 weeks (Control-Intervention Group). Intervention: POC BG (standard of care) uses commercially-available glucose meters for blood glucose monitoring. It is approved to be used in dialysis populations.
  Diagnostic Test: CGM will be used to collect outcomes variables during each phase (including during the POC BG testing).
Arm/Group | Real-time Dexcom CGM | Professional Dexcom CGM (Blinded)
Number analyzed (Participants) | 39 | 39
percentage of time in target range | 63.69 (23.58) | 54.24 (22.25)

3. Secondary Outcome: Mean % Time in Hypoglycemia (< 54 mg/dL)
Description: % time in hypoglycemia (<54 mg/dL) during the intervention phase in both groups (i.e. Real-time Dexcom CGM During CGM Intervention vs. Professional Dexcom CGM During Point-of-Care Glucose Intervention), as measured by CGM.
Time Frame: 8 weeks (after completion of both phases)
Population: Population analyzed per group included patients with usable data.
Measure: Mean (Standard Deviation); unit: percentage of time in hypoglycemia
Arm/Group | Real-time Dexcom CGM | Professional Dexcom CGM (Blinded)
Number analyzed (Participants) | 39 | 39
percentage of time in hypoglycemia | 0.46 (1.26) | 0.55 (2.10)

4. Secondary Outcome: % Time in Hyperglycemia (>180 mg/dL)
Description: % time in hyperglycemia (>180 mg/dL) during the intervention phase in both groups.(i.e. Real-time Dexcom CGM During CGM Intervention vs. Professional Dexcom CGM During Point-of-Care Glucose Intervention), as measured by CGM.
Time Frame: 8 weeks (after completion of both phases)
Population: Population analyzed per group included patients with usable data.
Measure: Mean (Standard Deviation); unit: percentage of time in hyperglycemia
Arm/Group | Real-time Dexcom CGM | Professional Dexcom CGM (Blinded)
Number analyzed (Participants) | 39 | 39
percentage of time in hyperglycemia | 35.07 (23.94) | 44.57 (22.90)

5. Secondary Outcome: % Time in Hyperglycemia (>250 mg/dl)
Description: % time in hyperglycemia (>250 mg/dL) during the intervention phase in both groups.(i.e. Real-time Dexcom CGM During CGM Intervention vs. Professional Dexcom CGM During Point-of-Care Glucose Intervention), as measured by CGM.
Time Frame: 8 weeks (after completion of both phases)
Population: Population analyzed per group included patients with usable data.
Measure: Mean (Standard Deviation); unit: percentage of time in hyperglycemia
Arm/Group | Real-time Dexcom CGM | Professional Dexcom CGM (Blinded)
Number analyzed (Participants) | 39 | 39
percentage of time in hyperglycemia | 13.18 (14.72) | 18.91 (18.76)

6. Secondary Outcome: Glycemic Variability [% Coefficient of Variation (%CV)
Description: % coefficient of variation will be measured during the intervention phase in both groups.(i.e. Real-time Dexcom CGM During CGM Intervention vs. Professional Dexcom CGM During Point-of-Care Glucose Intervention), as measured by CGM.
Time Frame: 8 weeks (after completion of both phases)
Population: Population analyzed per group included patients with usable data.
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variation
Arm/Group | Real-time Dexcom CGM | Professional Dexcom CGM (Blinded)
Number analyzed (Participants) | 39 | 39
percentage of coefficient of variation | 0.30 (0.05) | 0.31 (0.05)

7. Secondary Outcome: Mean Amplitude of Glucose Excursions (MAGE)
Description: Mean amplitude of glucose excursions (MAGE) will be measured during the intervention phase in both groups.(i.e. Real-time Dexcom CGM During CGM Intervention vs. Professional Dexcom CGM During Point-of-Care Glucose Intervention), as measured by CGM.
Time Frame: 8 weeks (after completion of both phases)
Population: Population analyzed per group included patients with usable data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Real-time Dexcom CGM | Professional Dexcom CGM (Blinded)
Number analyzed (Participants) | 39 | 39
mg/dL | 71.45 (19.71) | 72.24 (18.63)

8. Secondary Outcome: HbA1C at 3 Months Follow up
Description: HbA1C at 3 months follow up from baseline. Data will be exported from the electronic medical records.
Time Frame: Baseline, 3 months post-intervention
Population: Per standard of care, HbA1c was not repeated during the RCT before the three-month follow-up of the study (it was not collected by the dialysis center).
Measure: Mean (Standard Deviation); unit: percent of RBCs with glycated hemoglobin
Groups:
- All Participants: Participants received either Real-time Dexcom CGM Intervention or POC-BG Intervention first, and then switch to the remaining intervention after a 2 week wash out period.
Arm/Group | All Participants
Number analyzed (Participants) | 53
percent of RBCs with glycated hemoglobin
  Baseline | 7.21 (1.66)
  3 months post-intervention: number analyzed (Participants) | 0

9. Secondary Outcome: Number of Hospitalization or Emergency Room Visits for Hypoglycemia
Description: Rate of hospitalization or emergency room (ER) visits for hypoglycemia will be recorded at baseline (including 1 year prior to the start of the study) and at 3 months post study intervention.
Time Frame: Baseline, 3 months post-intervention
Population: Participants did not stay in the study for 3 months. Hence, data at 3 months was not possible to be collected by the dialysis center.
Measure: Number; unit: number of events
Arm/Group | All Participants
Number analyzed (Participants) | 53
number of events
  Number of hospitalization and emergency room visits for hypoglycemia at baseline | 21
  Number of hospitalization and emergency room visits for hypoglycemia at 3 months post-intervention: number analyzed (Participants) | 0

10. Secondary Outcome: Number of Hospitalization or Emergency Room Visits for Diabetes Ketoacidosis (DKA)
Description: Rate of hospitalization or emergency room visits for diabetes ketoacidosis will be recorded at baseline (including 1 year prior to the start of the study) and at 3 months post study intervention.
Time Frame: Baseline, 3 months post-intervention
Population: as for outcome 9
Measure: Number; unit: events
Arm/Group | All Participants
Number analyzed (Participants) | 53
events
  Number of hospitalization or emergency room visits for DKA at Baseline | 4
  Number of hospitalization or emergency room visits for DKA at 3 months post-intervention: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2.5 months
Groups:
- Real-time Dexcom CGM: Patients with type 2 DM treated with insulin and receiving hemodialysis used a real-time/personal CGM for 4 weeks
- Professional Dexcom CGM (Blinded): Patients with type 2 DM treated with insulin and receiving hemodialysis used POC BG for 4 weeks
Arm/Group | Real-time Dexcom CGM | Professional Dexcom CGM (Blinded)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 4/39 | 4/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real-time Dexcom CGM (N=39) | Professional Dexcom CGM (Blinded) (N=39)
Symptomatic Hypoglycemia <70mg/dl (Endocrine disorders) | 4 (14) | 4 (11)
Symptomatic Hypoglycemia <54mg/dl (Endocrine disorders) | 3 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT04473430/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT04473430/ICF_000.pdf